CLINICAL TRIAL: NCT05050188
Title: A Phase I, Randomized, Double-blind, Placebo- and Positive-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics/Pharmacodynamics (PK/PD) of Multiple Oral Doses of H008 (Carenoprazan Hydrochloride Tablets) in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics/Pharmacodynamics of Oral Doses of H008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Carephar Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KFP-2020-H008-HW-101
Record Dates: First submitted 2021-06-09; First posted 2021-09-20 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — 1-(5-(1H-indol-5-yl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Intervention Model Description: Two dose levels of H008 at 20 mg and 40 mg will be studied in two sequential cohorts. Each cohort will be enrolled with 12 subjects (8 on H008, 2 on placebo and 2 on positive control drug). Subjects are only allowed to participate in one of the two cohorts. Dose escalation to the next cohort will be permitted only when safety data until follow-up and PK data until 48 hours post-last dose, from all subjects in previous cohorts are reviewed, and the investigational product is deemed well tolerated.
Who Masked: Participant, Investigator
Masking Description: Both the investigational product and placebo will be given in a double blinded manner, while the positive control drug will be given in an open-label manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- cohort 1: H008 20mg (Experimental): H008 20mg tablets, orally, once, daily, for 7 days
  Interventions: Drug: H008
- cohort 1: H008 placebo 20mg (Experimental): H008 placebo 20mg tablets, orally, once, daily, for 7 days
  Interventions: Drug: H008 placebo
- cohort 1: Lansoprazole 30mg (Experimental): Lansoprazole 30mg capsule, orally, once, daily, for 7 days
  Interventions: Drug: Lansoprazole
- cohort 2: H008 40mg (Experimental): H008 40mg tablets, orally, once, daily, for 7 days
  Interventions: Drug: H008
- cohort 2: H008 placebo 40mg (Experimental): H008 placebo 40mg tablets, orally, once, daily, for 7 days
  Interventions: Drug: H008 placebo
- cohort 2: Lansoprazole 30mg (Experimental): Lansoprazole 30mg capsule, orally, once, daily, for 7 days
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: H008 — Drug administration after a minimum 10-hour overnight fasting. Subjects will be instructed to take the drugs with approximately 240 ml (8 oz) room temperature water.
  Arms: cohort 1: H008 20mg; cohort 2: H008 40mg
Drug: H008 placebo — Drug administration after a minimum 10-hour overnight fasting. Subjects will be instructed to take the drugs with approximately 240 ml (8 oz) room temperature water
  Arms: cohort 1: H008 placebo 20mg; cohort 2: H008 placebo 40mg
Drug: Lansoprazole — Drug administration after a minimum 10-hour overnight fasting. Subjects will be instructed to take the drugs with approximately 240 ml (8 oz) room temperature water
  Arms: cohort 1: Lansoprazole 30mg; cohort 2: Lansoprazole 30mg

SUMMARY:
This will be a Phase I, randomized, double-blind, positive- and placebo-controlled study to evaluate the safety, tolerability, and PK/PD of multiple oral doses of H008 in healthy adult subjects.

Two dose levels of H008 at 20 mg and 40 mg will be studied in two sequential cohorts. Each cohort will be enrolled with 12 subjects (8 on H008, 2 on placebo and 2 on positive control drug). Subjects are only allowed to participate in one of the two cohorts. Both the investigational product and placebo will be given in a double blinded manner, while the positive control drug will be given in an open-label manner.Dose escalation to the next cohort will be permitted only when safety data until follow-up and PK data until 48 hours post-last dose, from all subjects in previous cohorts are reviewed, and the investigational product is deemed well tolerated.

The study will consist of a screening period, a baseline period, a 7-day repeated-dose period and a safety follow-up period.

DETAILED DESCRIPTION:
Screening Period

After signing the informed consent, all subjects will undergo a screening assessment within 4 weeks prior to the start of study treatment (Days -28 to -3).

Baseline Period

Eligible subjects at screening will come to the clinic 2 days prior to the first dosing and begin their 11-day confinement period (Day -2 to Day 9). On Day -2, subjects will undergo baseline examinations. On Day -1, subjects will be monitored for their intragastric pH using a pH probe inserted into the stomach. The intragastric pH will be measured continuously for 48 h (Day -1 to Day 2), and data within the first 24 h will be used as baseline for PD evaluation. Subject's eligibility will be confirmed prior to first dosing (morning of Day 1).

Repeated-dose Period On each day during the treatment period, subjects will receive the investigational product (H008, 20 mg or 40 mg), matching placebos or positive control drug (Lansoprazole, 30 mg) according to the randomization schedule after a minimum 10-hour overnight fasting. No water is allowed within 1 hour before the drug administration. Subjects will be instructed to take the drugs with approximately 240 mL (8 oz) room temperature water, and swallow the tablets or capsules whole without chewing. On Days 1 to 7, no food or water is allowed within at least 2 hours post-dose, except the water ingested during dosing. Subjects should avoid lying down for 2 hours post-dose, except when ECG or vital sign measurements are performed. Standard lunch and dinner will be provided at approximately 4 and 10 hours post-dose on Days 1 and 7. On Days 2 to 6, standard breakfast, lunch and dinner will be provided at approximately 2, 5 and, 10 hours post-dose.

Serial PK blood samples will be collected for all subjects from pre-dose (Day 1) to 48 h after the last dose (Day 9). Detailed PK sampling plan is presented in Table 1.3-1. Another 24-h intragastric pH measurement will be performed from pre-dose on Day 7 until 24 h after the Day 7 dosing. All subjects will be closely monitored for safety during their stay in the clinic. Subjects will be discharged 48 hours after their last dosing (Day 9) if no clinically significant adverse events occur.

Follow-up Period

A follow-up safety assessment will be performed on Day 16 ± 1 at clinic. Unscheduled follow-ups should be performed for any clinically significant AE until it returns to normal or baseline or steady state.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male and female volunteers, 18 to 55 years of age, inclusive, at the time of dosing.
2. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the subject prior to any study-specific procedures).
3. Willingness and ability to comply with study procedures and follow-up examination.
4. Body mass index (BMI) ≥18 to ≤30 kg/m2 and total body weight ≥50.0 kg for males and ≥45.0 kg for females at screening.

   * If female and of childbearing potential (premenopausal and not surgically sterile), the subject:Must have a negative serum pregnancy test at screening. The serum pregnancy test must be obtained prior to the first administration of H-008 (≤72 hours prior to dosing) in all women.
   * Must agree to use an acceptable method of effective contraception for the duration of the study and for 3 months after receiving the last dose of study treatment.

   If male, the subject agrees to:
   * Use an acceptable method of effective contraception (a dual method of contraception: condom with spermicide in conjunction with use of an intrauterine device (IUD), condom with spermicide in conjunction with use of a diaphragm, condom with birth control patch or vaginal ring, or condom with oral, injectable, or implanted contraceptive) for the duration of the study and for 3 months after receiving study treatment.
   * Abstain from sperm donation for the duration of the study and for 90 days after receiving the last dose of study treatment.
   * Ensure their partner not get pregnant until 3 months following administration of the last dose of study treatment.
   * Be vasectomized for at least 6 months or take appropriate precautions to avoid fathering a child.
   * Male subjects who do not have sexual partners, they need to agree to remain abstinent at the time of screening, or agree to use a double barrier if they become sexually active.

   Use of hormonal contraceptive methods will not be allowed.
5. Medically healthy on the basis of medical history, and physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), as determined by the Investigator at Screening and each Check-In visit.
6. Medically healthy based on the absence of clinically significant abnormal vital sign measurements, clinical laboratory test results (especially tests for renal and hepatic function) as determined by the Investigator at Screening and Check-In visit.
7. Medically healthy based on the absence of clinically significant abnormal vital sign measurements, clinical laboratory test results (especially tests for renal and hepatic function) as determined by the Investigator at Screening and each Check-In visit.
8. Non-smokers (including nicotine-containing products) for at least 3 continuous months prior to the first dose.

Exclusion Criteria:

A subject is not eligible for the study if any of the following criteria is met:

1. Subjects who have a history of drug allergy or atopic allergic disease (e.g. asthma, urticaria, eczema, dermatitis, etc.) that were clinically significant, or allergic to any known ingredients and excipients of H008 and other PPIs drugs (e.g., Omeprazole, Lansoprazole, Ilaprazole, Esomeprazole, Rabeprazole, etc.).
2. History of alcohol or drug/substance abuse (within 2 years).
3. Positive urine drug screen or alcohol breath test at screening or baseline (Day -2).
4. Subjects who have history of unexplained syncope or fainting or a condition that predisposes them to syncope, such as hypotension, orthostatic hypotension, bradycardia or dehydration.
5. Subjects determined by the Investigator to have any medical condition that could jeopardize their health or prejudice study results (e.g., history of surgery of the gastrointestinal tract, which may interfere with absorption, except for appendectomy and cholecystectomy).
6. Subjects who have used P-gp and/or CYP 450 hepatic microsomal enzyme-inducing or inhibiting drugs (e.g., propafenone, voriconazole, fluconazole, cimetidine) within 30 days of first dosing.
7. Subjects with history or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychiatric disease, or active sexually transmitted disease.
8. History or clinical evidence of achlorhydria, severe gastrointestinal disease, particularly diarrhea or other conditions affecting gastrointestinal mobility or absorption.
9. Subjects who have difficulty in swallowing oral tablets or capsules.
10. History or presence of significant cardiovascular abnormalities, including without limitation, severe bradycardia, sick sinus syndrome, second- or third-degree atrial ventricular block, long QT syndrome, cardiogenic shock, and decompensated heart failure.
11. History or presence of pro-arrhythmic conditions, including a marked baseline prolongation of QTcF interval (i.e., repeated demonstration of a QTcF interval >450 milliseconds for males and >470 milliseconds for females) or a history of additional significant risk factors for torsade de pointes (e.g., family history of long QT syndrome), including any evidence of QTcF prolongation at screening;
12. Subjects who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody.
13. Subject is unable to refrain from or anticipated the use of any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [hypericum perforatum]), or grapefruits, grapefruit juice, blood oranges, apples and mulberry juice as well as vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard greens) beginning approximately 2 weeks prior to administration of the initial dose of investigational product, throughout the study, until the poststudy visit. Use of hormonal contraceptive methods will not be allowed.
14. Subjects donated blood (excluding plasma donation) of approximately 500 mL within 56 days prior to first dosing or donated plasma within 7 days prior to first dosing. Subjects will be advised not to donate plasma for 14 days after completing the study.
15. Subject consumes excessive amounts of caffeine for one month prior to investigational product administration, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.
16. Subjects who have participated in any other clinical trial within 30 days prior to the screening or five half lives of the investigational product received in the other trial.
17. Females who are pregnant, lactating, or likely to become pregnant during the study.
18. Abnormal gastric pH rhythms over 12 hours on Day -1, including abnormal pH increase lasting for more than 1 hour during non-eating or supine period, as judged by the physician.
19. Other conditions that an Investigator believes are not suitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
The number and incidence of AEs in HVs of multiple oral dose of H008 (Safety and Tolerability) | Up to final follow-up (Day16) or early termination.
  AEs
The number and incidence of subjects with clinically significant changes of physical examinations (Safety and Tolerability) | Baseline up to Day 16
  A baseline physical examination (defined as the pretreatment assessment immediately prior to the start of study drug) will consist of the following body systems: eyes、ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. All subsequent physical examinations should assess clinically significant changes from the baseline examination.
The number and incidence of subjects with abnormal vital signs of multiple oral dose of H008 (Safety and Tolerability) | Baseline up to Day 16
  Subjects with vital signs included body temperature(℃), blood pressure (both systolic and diastolic blood pressure ,mmHg), heart rate（beat per minute,BMP）, and respiratory rate (beat per minute,BMP）.
The number and incidence of subjects with clinical defined abnormal laboratory tests of multiple oral dose of H008 (Safety and Tolerability) | Baseline up to Day 16
  hematology，blood chemistry,urinalysis
The number and incidence of subjects with clinical defined abnormal of 12-lead ECG multiple oral dose of H008 (Safety and Tolerability) | Baseline up to Day 16
  Full 12-lead ECGs will be recorded using an ECG machine that automatically calculates the heart rate and measures HR、RR、PR, QRS, QT, QTc intervals. The investigator or other qualified physician will interpret each ECG using one of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.

SECONDARY OUTCOMES:
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  AUC0-t.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  AUC0-tau.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  AUC0-inf (if feasible).
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Cmax.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Ctroughs.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Tmax.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Kel.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  T1/2.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  CL/F.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Vd/F.
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Accumulation index (with steady state dosing).
To characterize the PK profiles of multiple oral doses of H008 in HVs. | through study completion,an average of 1 year
  Peak/trough fluctuation after single and multiple oral doses of H008.
Percentage of Time the pH is Greater than pH 3, pH 4 and pH 5 over a 24 Hour Period | Using a calibrated gastric pH monitor, the measurement of stomach pH will be made continuously over a 24-hour period at Baseline and over a 24-hour period following the administration of study on Days 1 and 7.
  Over a 24-hour period at Baseline and over a 24-hour period following the administration of study on Days 1 and 7
Percentage of Time the PH is Greater than pH 3, pH 4 and pH 5 from 8 PM to 8 AM | Using a calibrated gastric pH monitor, the measurement of stomach pH will be made continuously over a 12-hour period from 8 PM to 8 AM to assess nocturnal pH
  Over a 12-hour period from 8 PM to 8 AM on Days 1 and 7

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardhan KD, Hawkey CJ, Long RG, Morgan AG, Wormsley KG, Moules IK, Brocklebank D. Lansoprazole versus ranitidine for the treatment of reflux oesophagitis. UK Lansoprazole Clinical Research Group. Aliment Pharmacol Ther. 1995 Apr;9(2):145-51. doi: 10.1111/j.1365-2036.1995.tb00363.x. PMID 7605854
- [Background] Cheng Y, Liu J, Tan X, Dai Y, Xie C, Li X, Lu Q, Kou F, Jiang H, Li J. Direct Comparison of the Efficacy and Safety of Vonoprazan Versus Proton-Pump Inhibitors for Gastroesophageal Reflux Disease: A Systematic Review and Meta-Analysis. Dig Dis Sci. 2021 Jan;66(1):19-28. doi: 10.1007/s10620-020-06141-5. Epub 2020 Feb 24. PMID 32095968
- [Background] Chiba N, De Gara CJ, Wilkinson JM, Hunt RH. Speed of healing and symptom relief in grade II to IV gastroesophageal reflux disease: a meta-analysis. Gastroenterology. 1997 Jun;112(6):1798-810. doi: 10.1053/gast.1997.v112.pm9178669.
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] Echizen H. The First-in-Class Potassium-Competitive Acid Blocker, Vonoprazan Fumarate: Pharmacokinetic and Pharmacodynamic Considerations. Clin Pharmacokinet. 2016 Apr;55(4):409-18. doi: 10.1007/s40262-015-0326-7. PMID 26369775
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Fass R. Erosive esophagitis and nonerosive reflux disease (NERD): comparison of epidemiologic, physiologic, and therapeutic characteristics. J Clin Gastroenterol. 2007 Feb;41(2):131-7. doi: 10.1097/01.mcg.0000225631.07039.6d. PMID 17245209
- [Background] Fujiwara Y, Arakawa T. Epidemiology and clinical characteristics of GERD in the Japanese population. J Gastroenterol. 2009;44(6):518-34. doi: 10.1007/s00535-009-0047-5. Epub 2009 Apr 14. PMID 19365600
- [Background] Furukawa N, Iwakiri R, Koyama T, Okamoto K, Yoshida T, Kashiwagi Y, Ohyama T, Noda T, Sakata H, Fujimoto K. Proportion of reflux esophagitis in 6010 Japanese adults: prospective evaluation by endoscopy. J Gastroenterol. 1999 Aug;34(4):441-4. doi: 10.1007/s005350050293. PMID 10452674
- [Background] Kusano M, Hashizume K, Ehara Y, Shimoyama Y, Kawamura O, Mori M. Size of hiatus hernia correlates with severity of kyphosis, not with obesity, in elderly Japanese women. J Clin Gastroenterol. 2008 Apr;42(4):345-50. doi: 10.1097/MCG.0b013e318037556c. PMID 18277907
- [Background] Maekawa T, Kinoshita Y, Okada A, Fukui H, Waki S, Hassan S, Matsushima Y, Kawanami C, Kishi K, Chiba T. Relationship between severity and symptoms of reflux oesophagitis in elderly patients in Japan. J Gastroenterol Hepatol. 1998 Sep;13(9):927-30. doi: 10.1111/j.1440-1746.1998.tb00763.x. PMID 9794192
- [Background] Parsons ME, Keeling DJ. Novel approaches to the pharmacological blockade of gastric acid secretion. Expert Opin Investig Drugs. 2005 Apr;14(4):411-21. doi: 10.1517/13543784.14.4.411. PMID 15882117
- [Background] Richter JE, Bochenek W. Oral pantoprazole for erosive esophagitis: a placebo-controlled, randomized clinical trial. Pantoprazole US GERD Study Group. Am J Gastroenterol. 2000 Nov;95(11):3071-80. doi: 10.1111/j.1572-0241.2000.03254.x. PMID 11095320
- [Background] Maradey-Romero C, Fass R. New and future drug development for gastroesophageal reflux disease. J Neurogastroenterol Motil. 2014 Jan;20(1):6-16. doi: 10.5056/jnm.2014.20.1.6. Epub 2013 Dec 30. PMID 24466441
- [Background] Sharma VK, Leontiadis GI, Howden CW. Meta-analysis of randomized controlled trials comparing standard clinical doses of omeprazole and lansoprazole in erosive oesophagitis. Aliment Pharmacol Ther. 2001 Feb;15(2):227-31. doi: 10.1046/j.1365-2036.2001.00904.x. PMID 11148442
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Yadlapati R, Dakhoul L, Pandolfino JE, Keswani RN. The Quality of Care for Gastroesophageal Reflux Disease. Dig Dis Sci. 2017 Mar;62(3):569-576. doi: 10.1007/s10620-016-4409-6. Epub 2016 Dec 27. PMID 28028689